CLINICAL TRIAL: NCT01564901
Title: A Prospective Observational Study to Assess the Impact of RoActemra® on the Use of Glucocorticoids in Patients With Rheumatoid Arthritis Treated With the Standard of Care.
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Patients With Rheumatoid Arthritis Treated With Glucocorticoids
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27904
Record Dates: First submitted 2012-02-16; First posted 2012-03-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, observational, multicenter study will assess the efficacy and safety of RoActemra/Actemra (tocilizumab) on the use of glucocorticoids in patients with moderate to severe rheumatoid arthritis and an inadequate response to previous disease-modifying antirheumatic drugs or anti-TNF. Data will be collected for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, over 18 years of age
* Patients with moderate to severe rheumatoid arthritis (RA)
* Patients on a stable dose of prednisone or equivalent (>/=7.5 mg/day) for at least 4 weeks before study inclusion

Exclusion Criteria:

* Patients previously treated with RoActemra/Actemra
* Any contraindication to RoActemra/Actemra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis and concomitant treatment with glucocorticoids
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on treatment with RoActemra/Actemra who achieve prednisone (or equivalent) dose reduction of </= 5mg/day | Week 36

SECONDARY OUTCOMES:
Change from baseline in glucocorticoid dose | Week 36
Change from baseline in corticosteroid dose | Week 36
Proportion of patients treated with RoActemra/Actemra who reach Week 36 with a reduced glucocorticoid dose | Week 36
Proportion of patients treated with RoActemra/Actemra not receiving glucocorticoids | Week 36
Proportion of concomitant disease-modifying anti-rheumatic drug (DMARD) use | Week 36
Proportion of patients with inadequate response to prior treatment with disease-modifying antirheumatic drugs at baseline, who reach a prednisone (or equivalent) dose reduction of </= 5 mg/day | Week 36
Proportion of patients with inadequate response to prior treatment with anti-TNF at baseline, who reach a glucocorticoid dose reduction of </= 5 mg/day | Week 36
Proportion of patients meeting the physician's recommendaitons for glucocorticoid dose reduction | Week 36
Percentage change in Disease Activity Score 28 (DAS28) | Week 36
Percentage change in Simplified Disease Activity Index (SDAI) score | Week 36
Safety: Incidence of adverse events | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Spain (12):
  - Vitoria-Gasteiz, Alava
  - Alicante, Alicante
  - Elche, Alicante
  - Palma de Mallorca, Balearic Islands
  - Donostia / San Sebastian, Guipuzcoa
  - Huesca, Huesca
  - León, Leon
  - Ponferrada, Leon
  - Salamanca, Salamanca
  - Alzira, Valencia
  - Valencia, Valencia
  - Bilbao, Vizcaya